CLINICAL TRIAL: NCT01293643
Title: A Phase 3b, Comparative and Randomized Study to Assess the Efficacy and Safety of an Intravaginal Ovule Combination of Ketoconazole and Clindamycin Compared With an Intravaginal Cream Combination of Tetracycline and Amphotericin B for the Treatment of Bacterial Vaginosis and Vaginal Candidiasis, Either Mixed or Isolated
Brief Title: A Study to Compare the Efficacy and Safety of a Combination of Ketoconazole and Clindamycin Compared to Tetracycline/Amphotericin B Combination Cream for the Treatment of Bacterial Vaginosis and Vaginal Candidiasis (P08077)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P08077; BR 001-09 (Other: Schering Study Number)
Record Dates: First submitted 2011-02-09; First posted 2011-02-10 (Estimated); Last update posted 2015-08-10 (Estimated); Status verified 2015-08

CONDITIONS: Vaginosis, Bacterial; Candidiasis, Vulvovaginal
MeSH Terms: conditions — Vaginosis, Bacterial; Candidiasis, Vulvovaginal | interventions — Clindamycin; Tetracycline

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- clindamycin/ketoconazole combination (Experimental)
  Interventions: Drug: 100 mg clindamycin /800 mg ketoconazole vaginal ovule
- tetracycline hydrochloride/amphotericin B combination (Active Comparator)
  Interventions: Drug: 100 mg tetracycline hydrochloride /50 mg amphotericin B cream

INTERVENTIONS:
Drug: 100 mg clindamycin /800 mg ketoconazole vaginal ovule — 1 vaginal ovule for 3 consecutive days
  Arms: clindamycin/ketoconazole combination
Drug: 100 mg tetracycline hydrochloride /50 mg amphotericin B cream — 1 applicator (4 g) full of cream intravaginally for 7 to 10 days
  Arms: tetracycline hydrochloride/amphotericin B combination

SUMMARY:
This is a study to compare the safety and efficacy of the use of a intravaginal ovule containing a combination of Ketoconazole and Clindamycin to the use of an intravaginal cream containing a combination Tetracycline and Amphotericin B for the treatment of bacterial vaginosis and/or mixed or isolated vaginal candidiasis.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of vaginal candidiasis
* No Trichomonas vaginalis or any other protozoa
* No clinical evidences of infection by Neisseria gonorrhoeae, Chlamydia trachomatis, or viral infections

Exclusion Criteria:

* Known sensitivity to the formula components
* Pregnant or nursing patients
* Any gynecological condition contraindicating the use of vaginal ovule or cream.
* Use of any other local or systemic bactericidal, anti-protozoa or antifungal agent within the 2 weeks prior to the study start or during it
* Presence of other sexually transmitted diseases (except from Candidal vaginitis).
* History of recurrent candidiasis (≥4 episodes per year)
* Use of intra-uterine device, spermicides, or diaphragms
* Has metabolic or immune disorder
* Has abnormal uterine bleeding

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 99 (Actual)
Dates: Start 2010-05; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Percentage of participants that obtain clinical cure | Baseline up to Day 10
Percentage of participants that obtain microbiological cure | Baseline up to Day 10